CLINICAL TRIAL: NCT01745835
Title: Comparison Between 2L Coolprep® and Combination of 1L Coolprep® and Bisacodyl as Bowel Preparation for Colonoscopy
Brief Title: Comparison Between 2L Coolprep® and Combination of 1L Coolprep® and Bisacodyl as Bowel Preparation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Coolprep study
Record Dates: First submitted 2012-11-27; First posted 2012-12-10 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2017-02

CONDITIONS: Healthy Person; Bowel Preparation Before Colonoscopy
MeSH Terms: interventions — Bisacodyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2L Coolprep® (Active Comparator)
  Interventions: Drug: 2L Coolprep®
- 1L Coolprep® and Bisacodyl (Experimental)
  Interventions: Drug: 1L Coolprep® and Bisacodyl

INTERVENTIONS:
Drug: 2L Coolprep® — * Compositions/1L : Sodium Chloride 2.691g Potassium Chloride 1.015g Anhydrous sodium sulfate 7.5g PEG 3350 100g ascorbic acid 4.7g sodium ascorbate 5.9g
  Other Names: 2L Coolprep® (TaeJoon Pharmaceuticals, Seoul, Korea)
  Arms: 2L Coolprep®
Drug: 1L Coolprep® and Bisacodyl — 1. Coolprep® (TaeJoon Pharmaceuticals, Seoul, Korea)
     * Compositions/1L : Sodium Chloride 2.691g Potassium Chloride 1.015g Anhydrous sodium sulfate 7.5g PEG 3350 100g ascorbic acid 4.7g sodium ascorbate 5.9g
  2. Dulcolax-S® (Boehringer Ingelheim ,Seoul, Korea) * composition /1 tablet : Bisacodyl 5mg, docusate sodium 16.75mg
  Other Names: 1. Coolprep® (TaeJoon Pharmaceuticals, Seoul, Korea) : 1L; 2. Dulcolax-S® (Boehringer Ingelheim ,Seoul, Korea) : 4 tablet
  Arms: 1L Coolprep® and Bisacodyl

SUMMARY:
comparison of the use of Colyte® (ascorbic acid mixed polyethylene glycol solution) in two-liter versus one-liter volume and pretreatment with bisacodyl for colonoscopy preparation.

ELIGIBILITY:
Inclusion Criteria:

* willing to consent/undergo necessary procedures
* between the age of 20 and 75 years
* healthy persons planning to have a colonoscopy

Exclusion Criteria:

* history of abdominal surgery except appendectomy
* inflammatory bowel disease
* clinically or laboratory-confirmed ileus (both functional and mechanical)
* malignancy
* clinically severe cerebrovascular, cardiovascular, kidney, liver or hematologic disease
* dementia, cognitive impairment
* the use of prokinetics, antispasmodics, antidiarrheal drugs, laxatives or neuroleptics in 2 weeks
* known sensitivity to the agents used
* Pregnancy, Lactating woman

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2013-01-30 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
Bowel cleansing scale | on the day of the colonoscopy
  using SNUH scale

SECONDARY OUTCOMES:
Bowel cleansing scale of Right/Transverse/Left colon | on the day of the colonoscopy
  also using SNUH scale

OTHER OUTCOMES:
Patient's compliance | on the day of the colonoscopy
  using questionnaires
Patient's acceptance | on the day of the colonoscopy
  using questionnare
Patient's satisfaction | on the day of the colonoscopy
  using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jong Pil Im, M.D.,Ph.D., Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, City, South Korea

REFERENCES:
- [Derived] Kwon JE, Lee JW, Im JP, Kim JW, Kim SH, Koh SJ, Kim BG, Lee KL, Kim SG, Kim JS, Jung HC. Comparable Efficacy of a 1-L PEG and Ascorbic Acid Solution Administered with Bisacodyl versus a 2-L PEG and Ascorbic Acid Solution for Colonoscopy Preparation: A Prospective, Randomized and Investigator-Blinded Trial. PLoS One. 2016 Sep 2;11(9):e0162051. doi: 10.1371/journal.pone.0162051. eCollection 2016. PMID 27588943